CLINICAL TRIAL: NCT01720095
Title: A 1 Year Randomized, Controlled, Open-Label Study of the Impact of Flexible Doses of Niacin (NIASPAN) as an Adjunct to Antipsychotic Medication in the Treatment of First Episode Psychosis
Brief Title: Niapsan as Add -on Therapy to Antipsychotic Treatment in First Episode Psychosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDHA_RS/2010-116; NCT01041053 (obsolete NCT alias)
Record Dates: First submitted 2012-10-24; First posted 2012-11-02 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2012-10

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — Niacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Niaspan (Experimental): these are the first episode psychosis patients that are randomized to receive niaspan
  Interventions: Drug: Niaspan
- healthy control (No Intervention): this is the group of healthy controls for cognitive outcome measures
- first episode control group (No Intervention): first episode psychosis patients who are randomized to no intervention

INTERVENTIONS:
Drug: Niaspan
  Arms: Niaspan

SUMMARY:
The purpose of this study is to help understand if by adding Niaspan FCT (study drug) to antipsychotic medications will it help maintain or improve cognitve functioning.

ELIGIBILITY:
Inclusion Criteria:

ALL SUBJECTS

1. Must understand the nature of the study, must provide written informed consent prior to the conduct of any study procedures/assessments and are willing/able to participate in study procedures/assessments as specified in this protocol.
2. Must be between the ages of 18 - 35

PATIENTS

1. Within one year of initial DSM 1V TR diagnosis of schizophreniform psychosis, schizophrenia, schizoaffective disorder or psychotic disorder NOS
2. Outpatients
3. Females of child bearing potential who have a negative serum pregnancy test prior to enrolment and agree to use a reliable method of birth control (use of oral contraceptives or Norplant; contraceptive injections; contraceptive patch; double barrier method; intrauterine devices; partner with vasectomy or abstinence) during the study and for one month following the last dose of study drug.

HEALTHY CONTROLS

1. Age-matched to experimental groups

Exclusion Criteria:

1. Due to their underlying mental disorder are considered by the investigator(s) to be unable to provide informed consent and/or unwilling or unable to participate in study procedures/assessments
2. Are judged by the investigator(s) (based on history, mental status examination or clinical impression) as being at significant risk of self-injurious/suicidal or violent/homicidal behaviour
3. Meet criteria for substance abuse or dependence (excluding nicotine and caffeine) as defined by DSM IV-TR at the time of screening and/or within the preceding 6 months
4. Have unstable medical, psychiatric, neurological or behavioural disorders that may interfere in the conduct or interpretation of the study.
5. Have a history of pre-existing liver dysfunction and/or at screening have abnormal liver function tests (ALT>2x upper limit of normal; AST>3x upper limit of normal; Bilirubin>1.5x upper limit of normal)
6. Have a past or current history of peptic ulcer, gout or bleeding problems
7. Have a past or current history of hypophosphatemia
8. Have a history of head injury resulting in loss of consciousness of > 5 minutes or other neurological disorder (e.g., seizures, stroke, MS)
9. Are currently taking a vitamin or nutritional supplement containing a dose of niacin/nicotinic acid above 100 mg/day.
10. Are currently receiving treatment with any of the following medications:

    1. Anticoagulants
    2. Statins
    3. Antihypertensives
11. Are currently receiving treatment for Type 1 or Type 2 diabetes
12. Have a history of allergic reactions to NIASPAN or any of its non-medicinal ingredients (methylcellulose, povidone, stearic acid), niacin or nicotinic acid
13. Are currently participating in any other investigational drug study
14. Are a professional or staff member affiliated with the Nova Scotia Early Psychosis Program or are an immediate family member defined as spouse, parent, child, sibling, grandparent or grandchild

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2009-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
standardized and experimental measures of attention, memory, and executive function. Measurement tools=MATRICS; DalCAB | change in cognitive function from baseline to 3, 6, and 12 months
  Outcomes will be measured by comparison of pre-treatment, post-treatment and twelve month

CONTACTS AND LOCATIONS:
Overall Officials: Heather I Milliken, MD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- NS Early Psychosis Program, Halifax, Nova Scotia, Canada